CLINICAL TRIAL: NCT06240559
Title: In-vivo Treatment Verification for HDR Brachytherapy Patients Using an External Imaging Panel
Brief Title: In Vivo Treatment Verification of Brachytherapy
Status: Recruiting | Type: Observational
Sponsor: Maastricht Radiation Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: Verification of brachytherapy
Record Dates: First submitted 2024-01-26; First posted 2024-02-05 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Brachytherapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Device: External imaging panel — The IP will be placed on the side of the treatment table and will acquire data during the whole treatment, which will be compared against information derived from the treatment plan. The IP based method can detect errors and information about motion and treatment uncertainties that are not currently available.

SUMMARY:
To acquire data during High Dose Rate (HDR) brachytherapy treatments aiming to track the brachytherapy source inside the patient verifying the delivery of the treatment plan.

Medical images (CT,MRI and US) combined with software developed by the investigator will be employed to predict the response of the Investigational product during the treatment and will be used as reference.The IP will be placed on the side of the treatment table and will acquire data during the whole treatment, which will be compared against information derived from the treatment plan. The IP based method can detect errors and information about motion and treatment uncertainties that are not currently available.

DETAILED DESCRIPTION:
Medical images (CT,MRI and US) combined with software developed by us will be employed to predict the response of the IP during the treatment and will be used as reference. The IP will be placed on the side of the treatment table and will acquire data during the whole treatment, which will be compared against information derived from the treatment plan. The IP based method can detect errors and information about motion and treatment uncertainties that are not currently available.

The IP will not change the workflow or be in contact with the patient since the panel will be placed on the side of a treatment table/bed at a safe distance from the patient. The data will be acquired automatically when radiation is detected and only two cables are necessary to power the system and collect the data. The cables will be placed in a convenient position together with the cables of the treatment table, not interfering with the clinical workflow. Clinical staff will not need to perform any extra actions during the whole process of the data acquisition.

The analysis of the data generated during the trial will be performed offline to avoid a possible interruption of the treatment due to any error (real or false) that may be detected using the system.

ELIGIBILITY:
Inclusion Criteria:

* Treatment site Gynaecology (Endometrium/Cervix) and prostate
* Treatment: HDR Brachytherapy
* Patient will be treated on CT Couch
* Mentally competent patient

Exclusion Criteria:

* Incapacitated patient

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The developed method is expected to work for all treatments sites. However, HDR gynecological and prostate treatments are our main interest since they are the most common HDR treatments at Maastro.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-02-29 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dwell times | 1 year
  Verify all relevant parameters of the HDR treatment plan during treatment delivery such as dwell times (time in seconds).
  Brachytherapy treatments are delivered using two parameters, the first parameter is dwell times (the duration the radioactive source stays in a dwell position, measured in seconds (s)). Our system measures dwell times, comparing them against expected values. Note that this parameter can be further used to derive other metrics, such as radiation dose distributions (units in Gray (Gy)), as defined by the TG-43 AAPM dose formalism.
Dwell position | 1 year
  Verify all relevant parameters of the HDR treatment plan during treatment delivery such as dwell positions (distance in (milli)meters).
  Brachytherapy treatments are delivered using two parameters, the second parameter is dwell positions (a location where the radioactive source should stop, defined in centimeters (cm)) Our system measures dwell positions, comparing them against expected values. Note that this parameter can be further used to derive other metrics, such as radiation dose distributions (units in Gray (Gy)), as defined by the TG-43 AAPM dose formalism.

CONTACTS AND LOCATIONS:
Overall Officials: Maaike Berbée, Principal Investigator — Radiotherapist
Locations (1):
- Maastro, Maastricht, Limburg, Netherlands

IPD SHARING:
Plan to Share IPD: No